CLINICAL TRIAL: NCT04088305
Title: Clinical Evaluation of a Vancomycin Dosage Strategy Based on a Serum Trough Concentration Model in Elderly Patients With Severe Pneumonia
Brief Title: Vancomycin Dosage Strategy Based on a Trough Concentration Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qingtao Zhou, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y75505-03
Record Dates: First submitted 2019-09-07; First posted 2019-09-12 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pneumonia, Staphylococcal
Keywords: pneumonia; vancomycin; trough concentration; elderly patients
MeSH Terms: conditions — Pneumonia, Staphylococcal; Pneumonia | interventions — Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients of study group will accept vancomycin strategies decided by a serum trough concentration model.
  Interventions: Drug: Individualized therapy
- Control group (No Intervention): Patients of control group will accept vancomycin dosages decided by attending physician.

INTERVENTIONS:
Drug: Individualized therapy — Dosage of Vancomycin decided by a serum trough concentration model, instead of decided by attending physician
  Other Names: Vancomycin
  Arms: Study group

SUMMARY:
Study design:

Allocation: Randomized Endpoint classification: Efficacy study Masking: Open label Primary purpose: Treatment Primary endpoint: Incidence of reaching the target serum trough concentration Secondary endpoint: Clinical efficiency, Antibiotic use, acute kidney injury.

DETAILED DESCRIPTION:
This is a prospective randomized control trial. There are two groups, study group and control group. Patients of study group accepted vancomycin strategies decided by a serum trough concentration model, and patients of control group accepted vancomycin dosage decided by attending physician. The primary endpoint is the incidence of reaching the target serum trough concentration, the secondary endpoint are clinical efficiency, antibiotic use and side effects such as acute kidney injury, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients with doubted or diagnosed Methicillin-resistant Staphylococcus aureus severe pneumonia, and need vancomycin treatment.
* Sixty years and older.

Exclusion Criteria:

* younger than 60 years old
* Accepted blood purification therapy
* Pregnancy
* Positive HIV antibody titre
* Had known or suspected tuberculosis or other infections caused by fungi at baseline.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of vancomycin therapeutic serum trough concentrations | before the fifth vancomycin dosage
  The proportion of patients with vancomycin serum trough concentrations reaching target concentrations (≥15mg/L)will be compared between study group and control group

SECONDARY OUTCOMES:
Clinical success rate | Seven days after vancomycin withdrawal.
  the proportion of patients with clinical success
Vancomycin doses | At the end of vancomycin therapy, an average of 10 days.
  Vancomycin daily doses and totally doses
Incidence of acute kidney injury | At the end of vancomycin treatment, an average of 10 days.
  The incidence of vancomycin-associated acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Qingtao Zhou, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospita, Beijing, Beijing Municipality, China